CLINICAL TRIAL: NCT01026961
Title: A Randomized, Crossover, Double-Blind Study To Evaluate The Safety Of An Association Of Phenylephrine Hydrochloride 10mg + Acetaminophen 500mg + Dimethindene Maleate 1 Mg Compared To Phenylephrine Hydrochloride 10mg In Healthy Volunteers
Brief Title: Safety of Phenylephrine Hydrochloride, Acetaminophen, Dimethindene Maleate Compared to Phenylephrine Hydrochloride Alone in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study is no longer required by Brazil health authority.
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Biociências S.A
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 381-A-101
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Heart Rate; Blood Pressure; Arrhythmias
Keywords: Safety; heart rate; systolic and diastolic blood pressure; arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac; Systolic Murmurs | interventions — Oxymetazoline; Dimethindene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenylephrine HCL/Acetaminophen/Dimethindene Maleate (Experimental): Phenylephrine HCL/Acetaminophen/Dimethindene Maleate
  Interventions: Drug: Phenylephrine HCL/Acetaminophen/Dimethindene Maleate
- Phenylephrine hydrochloride (Active Comparator): Phenylephrine hydrochloride 10mg
  Interventions: Drug: Phenylephrine HCL

INTERVENTIONS:
Drug: Phenylephrine HCL — Phenylephrine HCL 10mg
  Arms: Phenylephrine hydrochloride
Drug: Phenylephrine HCL/Acetaminophen/Dimethindene Maleate — Phenylephrine HCL 10mg/Acetaminophen 500mg/Dimethindene Maleate 1mg
  Arms: Phenylephrine HCL/Acetaminophen/Dimethindene Maleate

SUMMARY:
This study will evaluate the safety of phenylephrine hydrochloride 10 mg + acetaminophen 500 mg + dimethindene maleate 1 mg compared to phenylephrine hydrocloride 10 mg alone in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 50 years;
* Clinical examination without abnormal findings
* Ability to understand the nature and purpose of the study, including the risks and adverse effects

Exclusion Criteria:

* Any cardiovascular disease, coronary artery disease, circulation problems or history of stroke, peripheral vascular disease or arrhythmia
* History of serious adverse reactions or hypersensitivity any drug
* Hypersensitivity to the drug study drugs or chemically related compounds

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
To compare the effect of phenylephrine hydrochloride 10mg + acetaminophen 500mg + dimethindene maleate 1mg and phenylephrine hydrochloride 10mg alone on vital signs | 15 days

SECONDARY OUTCOMES:
Electrocardiographic (ECG) monitoring and evaluation of heart rhythm following dosing | 15 days
To report and evaluate adverse events | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Biociências S.A, Study Director — Novartis
Locations (1):
- Scentryphar Pesquisa Clinica Ltda., Campinas, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://prsinfo.clinicaltrials.gov